CLINICAL TRIAL: NCT06587529
Title: Rigorous Evaluation of the READY to Stand Curriculum as a Tool to Prevent the Commercial Sexual Exploitation of Children Among Racially and Ethnically Diverse Urban Youth (PHASE III: Quasi Experimental Trial)
Brief Title: Rigorous Evaluation of the READY to Stand Curriculum to Prevent the Commercial Sexual Exploitation of Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katie M Edwards, Professor, School of Social Work, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23657
Record Dates: First submitted 2024-07-29; First posted 2024-09-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sex Trafficking; Sex Crimes; Commercial Sex; Sexual Violence; Child Abuse, Sexual; Sex Offense
Keywords: Human Trafficking; Sex Trafficking; Sex Crimes; Commercial Sex; Commercial Sexual Exploitation of Children; Prevention
MeSH Terms: conditions — Sex Work; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): READY to Stand© curriculum
  Interventions: Behavioral: The Set Me Free Project's (SMFP) READY to Stand (RTS)© Curriculum
- Control (No Intervention): control

INTERVENTIONS:
Behavioral: The Set Me Free Project's (SMFP) READY to Stand (RTS)© Curriculum — Students will receive the Ready to Stand (RTS)© programming over six school days, spread over six weeks. The program is delivered in mixed-gender groups of 20 to 40 students and includes videos, small and large group discussions, activities, worksheets, and ample opportunities for skill-building. This curriculum is intended to be one piece of comprehensive prevention strategies that has the potential to make immediate and sustained impacts on reducing rates of CSEC perpetration in the lives of youth, including those most vulnerable to this pernicious crime.
  Other Names: RTS©
  Arms: Treatment

SUMMARY:
The overall goal of the five-year project is to conduct both a process and rigorous outcome evaluation of The Set Me Free Project (SMFP)'s READY to Stand (RTS)© curriculum with an eye toward widespread dissemination to other U.S. communities, if deemed effective. Broadly, the investigators seek to determine the effect participation has on students: reductions in commercial sexual exploitation of children (CSEC) perpetration (the primary outcome); reductions in CSEC victimization, teen dating violence (TDV), and sexual violence victimization and perpetration; as well as increases in bystander intervention in CSEC situations compared to participants in the control condition (secondary outcomes).

DETAILED DESCRIPTION:
The commercial sexual exploitation of children (CSEC) is a public health crisis in the United States. Research has documented risk and protective factors across the social ecology for CSEC, that many perpetrators (traffickers, clients, recruiters) of CSEC are peers (e.g., romantic partners) and adolescents report opportunities to intervene in situations of peer victimization (although not necessarily specific to CSEC). Prevention efforts with adolescents that seek to (1) reduce risk for CSEC perpetration; (2) reduce risk for CSEC victimization; and (3) increase positive bystander intervention in situations of CSEC is urgently needed. Thus, the goal of this multi-stakeholder collaboration-which includes researchers, educators, practitioners, and youth-is to conduct both a process and rigorous outcome evaluation of The Set Me Free Project© (SMFP)'s READY to Stand (RTS)© curriculum-with an eye toward widespread dissemination to other U.S. communities, if deemed effective.

The RTS programming is for both students and school personnel. Student programming includes six, 45-minute modules implemented to high school students in mixed gender groups of ~25 students and provides students with CSEC psychoeducation, healthy relationship skills, identification of safe people, bystander intervention in CSEC situations, shifting school norms to be intolerant of all forms of violence, and valuing of self and others. School personnel participate in a training to equip them with skills to effectively respond to students' disclosures of CSEC, enhance cultural humility, and reinforce programming messages. Despite its potential for reducing CSEC, the RTS© has never been evaluated.

The investigators will conduct a quasi-experimental design study in which four traditional high schools and two alternative high schools (not including the two high schools that participated in NCT05988398) are assigned to treatment or control conditions. Students enrolled in spring elective courses (e.g., healthy relationships, psychology) in the four traditional high schools and all students in the two alternative high schools (n=3,218 [enrolled]) will complete baseline and immediate post, 6-, 12-, and 18-month follow-up surveys to test the hypothesis that participation in the RTS© program will lead to reductions in CSEC perpetration (primary outcome), as well as reductions in CSEC victimization and teen dating violence (TDV) and sexual violence victimization and perpetration, and increases in bystander intervention in CSEC situations compared to participants in the control condition (secondary outcomes) (Aim 2a). The investigators will assess mediators and demographic moderators of program impact (Aim 2b). Document via program observations of student and school personnel programming (Aim 2c), post-session surveys (n=1,459 students [enrolled in treatment schools]; n=150 school personnel [enrolled in treatment schools]) (Aim 2d), and post program implementation of key informant and stakeholder interviews (n=40: program facilitators [n=10], students [n=20], school personnel [n=10]) (Aim 2e) variations in implementation, unanticipated challenges, lessons learned, and perceptions of program impact. Determine costs associated with the program implementation (both student and school personnel programming) to inform future economic evaluation of the RTS (Aim 2f).

ELIGIBILITY:
Inclusion Criteria:

* enrolled in in Grade 9, 10, 11, or 12 at one of the eligible schools in the district
* able to understand spoken English

Exclusion Criteria:

• enrolled in either of the two schools involved in the corresponding Open Pilot Trial (NCT05988398)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3218 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Commercial Sexual Exploitation of Children (CSEC)-Victimization Experiences | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to assess students' self-reports of commercial sexual exploitation of children (CSEC) victimization; answers are binary (Yes/No) with an option not to answer. Scale information: items are summed and used to create two variables, one indicating if a student has ever experienced these activities and the other indicating if a student has experienced these activities in the past month. Higher scores indicate worse outcomes.
Commercial Sexual Exploitation of Children (CSEC)-Perpetration Experiences | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to assess students' self-reports of commercial sexual exploitation of children (CSEC) victimization perpetration; answers are binary (Yes/No) with an option not to answer. Scale information: items are summed and used to create two variables, one indicating if a student has ever experienced these activities and the other indicating if a student has experienced these activities in the past 1 or 6 months (1-month time frame utilized at baseline, 6-month time frame utilized for all follow ups). Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Commercial Sexual Exploitation of Children (CSEC)-Bystander Opportunity and Action | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Response options range from 0 to "10 or more" with an option to not answer. If participants report "one or more times" they are then asked how many times they took the specified actions. Eleven actions are listed, two of which are negative behaviors, such as doing nothing, with the other nine actions being positive behaviors, such as trying to stop the situation. For each positive action, students' responses are re-coded into a binary variable where 0=did not take action and 1=did take action. For each negative item, responses are reverse-scored. Items are then summed to create an overall score that could range from 2 to 7, with a higher score indicating better outcomes.
Sexual Assault | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to assess students' self-reports of experiencing sexual assault victimization and perpetration; answers are binary (Yes/No) with an option not to answer. Items are summed, with higher scores indicating worse outcomes.
Sexual Harassment | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to assess students' self-reports of experiencing sexual harassment victimization and perpetration; answers are binary (Yes/No) with an option not to answer. Items are summed, with higher scores indicating worse outcomes.
Stalking | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to assess students' self-reports of experiencing stalking victimization and perpetration; answers are binary (Yes/No) with an option not to answer. Items are summed, with higher scores indicating worse outcomes.
Dating Violence (MARSHA) | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items to the Measure of Adolescent Relationship Harassment and Abuse (MARSHA) will be used to assess dating violence victimization and perpetration. Each subscale was summed so that higher scores indicate higher frequencies of Intimate Partner Violence (IPV), a worse outcome. Each subscale is also dichotomized to represent the absence or presence of that type of IPV.
Youth Violence | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Behaviorally worded items from the Youth Risk Behavior Surveillance System (YRBSS) will be used to measure physical fights, fear of going to school, and weapon carrying; answers are binary (Yes/No) with an option not to answer. Items are summed, with higher scores indicating worse outcomes.
Depression | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  The Patient Health Questionnaire (PHQ-9) modified will be used to measure depression; items are rated from 0 ("Not at all") to 3 ("Nearly every day"). Higher scores indicate higher depressive symptomology, a worse outcome.
Alcohol Use | Time 1 (baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Items from Monitoring the Future will be used to measure past month alcohol use and alcohol intoxication; items are rated from 0 ("0 times") to 9 ("40+ times"), with higher scores indicating worse outcomes.
Academic and Career Commitment | Time 1 (baseline), Time 2 (approximately three months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Items to measure students' intentions on graduating high school/getting a GED as well as having a job/career, rated from 1 ("not true at all of me") to 4 ("extremely true of me"), with an option not to answer. A total score is calculated by taking the average of the five items, with higher scores indicating better outcomes.

OTHER OUTCOMES:
Commercial Sexual Exploitation of Children (CSEC) Knowledge | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Researcher created items to assess knowledge about sex trafficking (that aligns with the student programming being received). This measure is comprised of 19 items across four subscales. For each subscale, a total score is calculated by taking the mean of the items. The mean is the proportion of items answered correctly; scores can range from 0-1, with a higher score indicating better outcomes.
Efficacy to Avoid Victimization (Efficacy) | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Researcher created items to assess confidence in resistance to being a victim of commercial sexual exploitation of children (CSEC). Answer options ranged from "not at all confident" (1), "somewhat confident" (2), to "very confident" (3), with an option not to answer. Items are summed with higher scores indicating better outcomes.
Valuing of Self and Others | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Researcher created items to assess the extent to which students value themselves and others. Items were created based on positive youth development and dignity literature. Items comprise two subscales, one on self-value and the next on the value of others, each with eight statements. Participants are asked to rate the statements on a scale from "strongly disagree" (1) to "strongly agree" (4). One item in each section was reverse coded. Scores for the subscales were calculated by taking the average of the subscale items, with higher scores indicating better outcomes.
Healthy Relationships Skills | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Items adapted from the Communications Skills Test and Sexual Communication Self-Efficacy Scale to assess conflict management and sexual refusal skills, used to assess students' communication skills with a romantic partner. In addition, two items were created by the researchers to assess consent and respecting boundaries that are based on the READY to Stand© program. Answer options included "very difficult" (1), "difficult" (2), "easy" (3), and "very easy" (4). Higher scale scores reflect healthier relationship communication skills, a better outcome.
Bystander Readiness to Help | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  The Denial Subscale of the Bystander Readiness to Help measure: participants rate five statements on a scale from "strongly disagree" (4) to "strongly agree" (1), with an option not to answer. The composite score is the mean of the five items, with higher scores indicating better outcomes.
Social Norms | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  This scale is composed of a series of statements that gauged personal beliefs, perceptions of friends, perceptions of other high school students in this district, and perceptions of school personnel in the district regarding their beliefs on sex trafficking. Participants rate statements on a scale from "strongly disagree" (1) to "strongly agree" (4), with an option not to answer. Items are summed, with higher scores indicating better outcomes.
Prevention Related Conversations with School Personnel | Time 1 (baseline), Time 2 (approximately 3 months post-baseline), Time 3 (six months post-baseline), Time 4 (twelve months post-baseline, Time 5 (eighteen months post-baseline)
  Items to assess conversations (from students' perspectives) with school personnel about healthy relationships, valuing self and others, healthy relationship skills, sex trafficking, dating violence, and bystander intervention; participants rate statements on a scale from "strongly disagree" (1) to "strongly agree" (4), with an option not to answer. Items are summed, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle Dalla, PhD, Study Director — University of Nebraska Lincoln; Lorey Wheeler, PhD, Study Director — University of Nebraska Lincoln; Katie Edwards, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- [school districts in the Midwest], Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The level of public access will be restricted such that the data set will be available under certain use restrictions. More specifically, the PI intends to share the aggregated, de-identified quantitative survey data if users commit to the following: (a) using the data only for research purposes and not to identify any individual participant; (b) securing the data using appropriate computer technology; and (c) destroying or returning the data after analyses are completed. If the researcher agrees, in writing, to these stipulations, the PI will send the approved researcher the dataset prepared using SPSS 27.0 (or the latest version available). The prepared data set will not include identifying information about participants, schools, or Des Moines Public Schools. Research participants will be identified by number. Schools will be coded as a number so as not to identify the participating schools/district.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available likely around fall 2027. It will be made available indefinitely.
Access Criteria: See above in Plan Description.

REFERENCES:
- [Background] Edwards KM, Banyard VL, Waterman EA, Mitchell KJ, Jones LM, Kollar LMM, Hopfauf S, Simon B. Evaluating the Impact of a Youth-Led Sexual Violence Prevention Program: Youth Leadership Retreat Outcomes. Prev Sci. 2022 Nov;23(8):1379-1393. doi: 10.1007/s11121-022-01343-x. Epub 2022 Mar 18. PMID 35303249
- [Background] Cook-Craig PG, Coker AL, Clear ER, Garcia LS, Bush HM, Brancato CJ, Williams CM, Fisher BS. Challenge and opportunity in evaluating a diffusion-based active bystanding prevention program: Green Dot in high schools. Violence Against Women. 2014 Oct;20(10):1179-202. doi: 10.1177/1077801214551288. Epub 2014 Sep 24. PMID 25255794
- [Background] Lipson, J. (2001). Hostile hallways: Bullying, teasing, and sexual harassment in school. AAUW Educational Foundation, 1111 Sixteenth Street, NW, Washington, DC 20036.
- [Background] Rothman EF, Paruk J, Cuevas CA, Temple JR, Gonzales K. The Development of the Measure of Adolescent Relationship Harassment and Abuse (MARSHA): Input From Black and Multiracial, Latinx, Native American, and LGBTQ+ Youth. J Interpers Violence. 2022 Mar;37(5-6):2126-2149. doi: 10.1177/0886260520936367. Epub 2020 Jul 5. PMID 32627640
- [Background] Centers for Disease Control and Prevention. 2019 Youth Risk Behavior Surveillance System results. U.S. Department of Health & Human Services. https://www.cdc.gov/healthyyouth/data/yrbs/index.htm
- [Background] Johnson JG, Harris ES, Spitzer RL, Williams JB. The patient health questionnaire for adolescents: validation of an instrument for the assessment of mental disorders among adolescent primary care patients. J Adolesc Health. 2002 Mar;30(3):196-204. doi: 10.1016/s1054-139x(01)00333-0. PMID 11869927
- [Background] Monitoring the future national survey results on drug use, 1975-2020: Overview, key findings on adolescent drug use. https://eric.ed.gov/?id=ED611736.
- [Background] Hulsey L., Zief, S., & Murphy, L. PREP Entry and Exit Survey Measures Guide. 2022. https://www.prepeval.com/DataCollection/50273%20Data%20Dictionary%202022.pdf
- [Background] Project SMF. READY to Stand Curriculum. 2021
- [Background] Ziebertz H-G, Döhnert S, Unser A. Predictors of attitudes towards human dignity: An empirical analysis among youth in Germany. Religion and civil human rights in empirical perspective. Springer; 2018:17-60.
- [Background] Lebech M. What is human dignity? Maynooth philosophical papers. 2004;2:59-69.
- [Background] Bal M. A Review of Human Dignity. Dignity in the Workplace. 2017:41-66.
- [Background] Bowers EP, Li Y, Kiely MK, Brittian A, Lerner JV, Lerner RM. The Five Cs model of positive youth development: a longitudinal analysis of confirmatory factor structure and measurement invariance. J Youth Adolesc. 2010 Jul;39(7):720-35. doi: 10.1007/s10964-010-9530-9. Epub 2010 Apr 16. PMID 20397040
- [Background] Park, N. (2004). Character strengths and positive youth development. The Annals of the American Academy of Political and Social Science, 591(1), 40-54.
- [Background] Lerner, R. M., Almerigi, J. B., Theokas, C., & Lerner, J. V. (2005). Positive youth development a view of the issues. The journal of early adolescence, 25(1), 10-16.
- [Background] Jenkins N, Saiz C. The communication skills test. Unpublished manuscript, University of Denver, Denver, CO. 1995
- [Background] Quinn-Nilas C, Milhausen RR, Breuer R, Bailey J, Pavlou M, DiClemente RJ, Wingood GM. Validation of the Sexual Communication Self-Efficacy Scale. Health Educ Behav. 2016 Apr;43(2):165-71. doi: 10.1177/1090198115598986. Epub 2015 Aug 17. PMID 26286296
- [Background] Edwards KM, Banyard VL, Sessarego SN, Stanley LR, Mitchell KJ, Eckstein RP, Rodenhizer KAE, Leyva PC. Measurement Tools to Assess Relationship Abuse and Sexual Assault Prevention Program Effectiveness Among Youth. Psychol Violence. 2018 Sep;8(5):537-545. doi: 10.1037/vio0000151. PMID 31660253
- [Background] Banyard VL. Measurement and correlates of prosocial bystander behavior: the case of interpersonal violence. Violence Vict. 2008;23(1):83-97. doi: 10.1891/0886-6708.23.1.83. PMID 18396583
- [Background] Waterman EA, Banyard VL, Edwards KM, Mauer VA. Youth perceptions of prevention norms and peer violence perpetration and victimization: A prospective analysis. Aggress Behav. 2022 Jul;48(4):402-417. doi: 10.1002/ab.22024. Epub 2022 Feb 16. PMID 35174509
- [Background] Edwards KM, Banyard VL, Kirkner A. Parents Matter: A Descriptive Study of Parental Discussions With Teens About Violence Prevention and Related Topics. J Interpers Violence. 2022 Apr;37(7-8):NP3856-NP3874. doi: 10.1177/0886260520949153. Epub 2020 Aug 26. PMID 32842824
- [Background] Edwards KM, Sessarego SN, Stanley LR, Mitchell KJ, Eckstein RP, Rodenhizer KAE, Leyva PC, Banyard VL. Development and Psychometrics of Instruments to Assess School Personnel's Bystander Action in Situations of Teen Relationship Abuse and Sexual Assault. J Interpers Violence. 2021 Feb;36(3-4):NP1586-1606NP. doi: 10.1177/0886260517746946. Epub 2017 Dec 20. PMID 29295034
- [Background] Monitoring the future national survey results on drug use, 1975-2020: Overview, key findings on adolescent drug use. https://eric.ed.gov/?id=ED611736
- [Background] Johnston, Lloyd D.; Miech, Richard A.; O'Malley, Patrick M.; Bachman, Jerald G.; Schulenberg, John E.; Patrick, Megan E. (2022) Demographic Subgroup Trends among Adolescents in the Use of Various Licit and Illicit Drugs, 1975-2021. Monitoring the Future Occasional Paper Series. Paper 97. Institute for Social Research.
- [Background] Franchino-Olsen H, Martin SL, Halpern CT, Preisser JS, Zimmer C, Shanahan M. Adolescent Experiences of Violence Victimizations Among Minors Who Exchange Sex/Experience Minor Sex Trafficking. J Interpers Violence. 2022 Sep;37(17-18):NP16277-NP16301. doi: 10.1177/08862605211021967. Epub 2021 Jun 30. PMID 34192962
- [Background] Rothman EF, Farrell A, Paruk J, Bright K, Bair-Merritt M, Preis SR. Evaluation of a Multi-Session Group Designed to Prevent Commercial Sexual Exploitation of Minors: The "My Life My Choice" Curriculum. J Interpers Violence. 2021 Oct;36(19-20):9143-9166. doi: 10.1177/0886260519865972. Epub 2019 Jul 27. PMID 31354019